CLINICAL TRIAL: NCT02583802
Title: The Clinical Study of Improving the Thirst and Hypotension of Hemodialysis Patients by Ear Pills Combined With Shengmai Capsule
Brief Title: The Clinical Study of Improving the Thirst and Hypotension of Hemodialysis Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: Wang Jing Hospital (Other); Beijing First Hospital of integrated Chinese and Western Medicine (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Cao po, Chief physician, Professor, master's tutor, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-ZYLC-003
Record Dates: First submitted 2015-10-13; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Intradialytic Hypotension
Keywords: MHD; ear pills; Shengmai capsule; Chinese medicine treatment
MeSH Terms: interventions — fructus schizandrae, radix ginseng, radix ophiopogonis drug combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group received regular hemodialysis treatment, no given Ear pills and Shengmai capsule completed in the treatment of the first stage. After 4 weeks after a washout period, two groups of cross accept the next phase of treatment.
- Ear pills and Shengmai capsule (Experimental): On regular hemodialysis based on given auricular Ear pills and Shengmai capsule
  Interventions: Drug: Ear pills; Drug: Shengmai capsule

INTERVENTIONS:
Drug: Ear pills — The clinical design of this study was a randomized crossover trial. This experiment research is divided into two stages, each stage is 8 weeks. After 4 weeks after a washout period, two groups of cross accept the next phase of treatment.
  Arms: Ear pills and Shengmai capsule
Drug: Shengmai capsule — The clinical design of this study was a randomized crossover trial. This experiment research is divided into two stages, each stage is 8 weeks.
  Arms: Ear pills and Shengmai capsule

SUMMARY:
This clinical study is to observe the improvement of MHD (maintenance hemodialysis) patients, quality of life，after applying therapy combining Auriculotherapy and Shengmai capsule. As a compliment to each other, Traditional Chinese Medicine and Modern Medicine form a joint and help improving life quality of MHD patients. Through the therapy, MHD patients, symptoms of thirst are improved, the incidence of intradialytic hypotension is reduced, the intake of water and sodium is lessen and the weight gain during dialysis is controlled, which consequently reduce cardiovascular and cerebrovascular complications and eventually reduce the mortality of MHD patients. Aiming to improve patients, thirst symptom and reduce the incidence of intradialytic hypotension, this study prospectively followed 144 MHD patients using multicenter prospective randomized crossover controlled clinical studies, using KT/V, URR, improvement of thirst, blood pressure and cognitive assessment as observational index. Multiple questionnaire surveys are conducted to understand patients, life quality from different angle. The use of Auriculotherapy is simple and effective and Shengmai capsule conforms to patients, syndrome, which is consistent with TCMs principle of "syndrome differentiation and treatment"and the theory of preventive treatment. The study not only expends the use of TMC in hemodialysis treatment, but also suggests a set of easy therapeutic schedules to improve the quality of life in patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
3.1 research object 3.1.1 case: 3.1.1.1 Beijing University of Chinese Medicine Dongzhimen hospital 48 cases 3.1.1.2 54 cases of Oriental Hospital of Beijing University of Chinese Medicine 3.1.1.3 Chinese Academy of traditional Chinese medicine, Wangjing Hospital, 20 cases 3.1.1.4 28 case of Beijing Pinggu Hospital of Traditional Chinese Medicine 3.1.2 diagnostic criteria: 3.1.2.1: syndrome score standard: according to the traditional Chinese medicine clinical research guiding principle (2002), chronic renal failure syndrome of deficiency of both qi and Yin compiled score table and determine the inclusion criteria.

Diagnostic criteria of hypotension in 3.1.2.2:

Referring to the Ministry of health of the people's Republic of China promulgated the "blood purification standard operating procedures (2010 Edition)" in the "blood dialysis hypotension prevention and control standards for the prevention and control of standard operating procedures", the diagnostic criteria are as follows: (1) can be diagnosed: (1) systolic blood pressure reduction of more than 20mmHg; (2) the average arterial pressure decreased more than 10mmHg.

3.1.2.3 mouth thirst intensity score The investigators will mouth thirst intensity score table (XQ) eight problems in the translation into Chinese questionnaire, each question by visual rating scale method and by the patients according to their own scoring. The higher score indicated the mouth thirst more serious or mouth thirst caused discomfort heavier, and the summation of the scores of each question and convert it to a range of 0 to 100 score, resulting score higher mouth thirst more serious degree.

3.1.4.2 on the treatment of Chinese and Western medicine treatment of poor compliance.

3.1.4.3 infection, fever, acute heart failure or diabetes and blood glucose control is not ideal.

3.1.4.4 for the preparation of the capsule and the skin allergic patients with adhesive tape.

3.1.4.5 patients can not cooperate or not sign the informed consent. 3.1.5 removing and dropping standard 3.1.5.1 all cases that are not included in the criteria for inclusion in the inclusion criteria shall be excluded; 3.1.5.2 clinical information is not the whole case to be removed. 3.2 case grouping method This research is to set up experimental group (Western medicine routine + acupoint therapy combined with birth control group) and the control group (Western medicine group). To meet the inclusion exclusion criteria of the subjects, using random number table method to produce random sequence number, according to the random sequence number to the subjects were assigned to different treatment groups.

3.3 treatment method and treatment The clinical design of this study was a randomized crossover trial. This experiment research is divided into two stages, each stage is 8 weeks. Experimental group on regular hemodialysis based on given auricular therapy selected export sympathetic endocrine, God door, massage time for about 1 minute, 3 ~ 5 times / day, each taking one side ear, 3 ~ 7 days take on the other side of the ear; Shengmai capsules and Shengmai Capsules (ChiaTai Qingchunbao Pharmaceutical Co., Ltd., Chinese medicine quasi word Z33021036, every grain of 0.3g. Ingredients: ginseng, ophiopogon root, Schisandra 3 capsules / time, 3 times / day. Control group received regular hemodialysis treatment, completed in the treatment of the first stage. After 4 weeks after a washout period, two groups of cross accept the next phase of treatment.

3.5 observation index 3.5.1 safety index: Into the group, crossover trial and the end of the experiment were used to detect the blood routine hemodialysis patients, before and after dialysis and renal ion, and serum albumin.

3.5.2 evaluation index:

1. and KT/V: and URR were measured in the clinical observation of the biochemical, dialysis, and body weight at the end of the biochemical, dialysis, and weight gain of hemodialysis and Improvement Center. URR = (BUN) /BUN (BUN = 100%) + (4 *) + (3.5 * R) * KT/V (R = R) (BUN = 0.03) (LN = UF/W) (BUN =).
2. thirst improvement: combined with clinical experience, thirst was divided into eight levels (combined with patients' self perception and thirst intensity score), making a thirst scale, in the group, when the end of the experiment and the end of the experiment, respectively, to observe the improvement of thirst before and after treatment.
3. on the basis of the analysis of the improvement of the low blood pressure (first): according to the diagnostic criteria of hypotension in hemodialysis patients, the incidence of hypotension in the experimental group and the second stage was compared with that of the experimental group and the control group.
4. the quality of life improvement in dialysis patients: in the clinical observation, the patients were treated with in-depth interviews, the use of key data extraction methods, to reflect the quality of life of patients with dialysis information; in the clinical observation of the patients, the cross exchange and the end of the life quality of SF-36 patients.

ELIGIBILITY:
Inclusion Criteria:

1. in the blood purification center hemodialysis (2-4 times / week, the same below) more than 3 months;
2. in line with the deficiency of both qi and Yin syndrome score greater than or equal to 9 points and thirsty XQ scores greater than or equal to 8 points; or deficiency of both qi and Yin syndrome score greater than or equal to 9 points and dialysis hypotension occurred frequency is greater than or equal to 1 / 5 of dialysis patients;
3. between 18-80, the condition is basically stable;
4. have better treatment compliance, signed informed consent.

Exclusion Criteria:

1. patients in the blood purification center of the law for less than 3 months.
2. the treatment of Chinese and Western medicine treatment of poor compliance.
3. infection, fever, acute heart failure or diabetes and blood glucose control is not ideal.
4. the patients with the capsule preparation and adhesive tape skin allergy.
5. patients unable to cooperate or not sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The measurement of blood pressure | 8 weeks
  According to the diagnostic criteria of hypotension in hemodialysis patients， To summarize the incidence of hypotension in the experimental group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Beijing University of Chinese Medicine Beijing University of Chinese Medicine, Principal Investigator — Chinese Ministry of Education
Locations (1):
- Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Eisbruch A, Kim HM, Terrell JE, Marsh LH, Dawson LA, Ship JA. Xerostomia and its predictors following parotid-sparing irradiation of head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Jul 1;50(3):695-704. doi: 10.1016/s0360-3016(01)01512-7. PMID 11395238
- [Background] Jabbari S, Kim HM, Feng M, Lin A, Tsien C, Elshaikh M, Terrel JE, Murdoch-Kinch C, Eisbruch A. Matched case-control study of quality of life and xerostomia after intensity-modulated radiotherapy or standard radiotherapy for head-and-neck cancer: initial report. Int J Radiat Oncol Biol Phys. 2005 Nov 1;63(3):725-31. doi: 10.1016/j.ijrobp.2005.02.045. PMID 16199308
- [Background] Lin A, Kim HM, Terrell JE, Dawson LA, Ship JA, Eisbruch A. Quality of life after parotid-sparing IMRT for head-and-neck cancer: a prospective longitudinal study. Int J Radiat Oncol Biol Phys. 2003 Sep 1;57(1):61-70. doi: 10.1016/s0360-3016(03)00361-4. PMID 12909216
- [Background] Pacholke HD, Amdur RJ, Morris CG, Li JG, Dempsey JF, Hinerman RW, Mendenhall WM. Late xerostomia after intensity-modulated radiation therapy versus conventional radiotherapy. Am J Clin Oncol. 2005 Aug;28(4):351-8. doi: 10.1097/01.coc.0000158826.88179.75. PMID 16062076